CLINICAL TRIAL: NCT02288390
Title: Oral Care as a Preventive Measure of VAP; Miswak Versus Chlorhexidine and Toothbrush, a Prospective, Randomized Controlled Study
Brief Title: Oral Care as a Preventive Measure of VAP; Miswak Versus Chlorhexidine and Toothbrush.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alexandria (Other)
Responsible Party: Principal Investigator, Ahmed M El-Mehalawy, Egypt, Alexandria, Sidi Gaber, University of Alexandria
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Faculty of Medicine 10.07.2007
Record Dates: First submitted 2014-10-31; First posted 2014-11-11 (Estimated); Last update posted 2014-11-11 (Estimated); Status verified 2014-11

CONDITIONS: Ventilator Associated Pneumonia
Keywords: VAP; Oral care; Chlorhexidine; Miswak (Sewak)
MeSH Terms: conditions — Pneumonia, Ventilator-Associated

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Miswak (Sewak) (Active Comparator): Miswak (sewak) oral care applied 4 hourly for oral care in mechanically ventilated patients.
  Interventions: Procedure: Oral care in mechanically ventilated patients
- Chlorhexidine/ toothbrush (Active Comparator): Chlorhexidine 0.12 % plus toothbrushing oral care applied 4 hourly for oral care in mechanically ventilated patients.
  Interventions: Procedure: Oral care in mechanically ventilated patients

INTERVENTIONS:
Procedure: Oral care in mechanically ventilated patients — Oral care comparing Chlorhexidine and toothbrush versus Miswak ( the twig of Arak, Salvadora perscia, tree)

SUMMARY:
Dental plaque score calculation and swabs of Oropharynx and teeth were collected on admission. For group I, Miswak stick was used 4 hourly for oral care. For group II, 0.12% Chlorhexidine/ toothbrush were used 4 hourly

DETAILED DESCRIPTION:
The selected patients were randomized into 2 groups by the conventional method of randomization. For each patient the following parameters were collected: patient data; age, gender; history of smoking; chronic health problems; history of drugs as steroids, chemotherapy, current antimicrobial therapy; and the primary cause of hospital and ICU admission and mechanical ventilation.

Clinical examination included assessment of disease severity on admission by Acute Physiology and Chronic Health Evaluation (APACHE II) scoring system, oral and dental examination, and dental plaque score calculation. Oropharyngeal and dental swabs were collected on admission.

The preventative VAP bundle was applied to all patients in both groups. For group I, Miswak was used for oral care, patient's teeth were brushed every 4 hours using a Miswak stick after scraping of half an inch bark from the stick end then Miswak tip was washed and compressed to make it brush like. Both buccal and lingual surfaces of teeth were brushed using mechanical method for plaque removal (in direction away from gingival margin,). The patient's tongue was brushed when possible and lip moisturizer was applied as needed. The brush like end of sewak stick was cut and replaced daily.

For group II, the patient's teeth were brushed every 4 hours using a soft toothbrush with 0.12% Chlorhexidine solution. Both buccal and lingual surfaces of teeth were brushed using mechanical method for plaque removal (in direction away from gingival margin,). The patient's tongue was brushed when possible and lip moisturizer was applied as needed. The toothbrush was boiled for one minute every day.

Patients in both groups were monitored for the efficacy of oral care in term of plaque score and halitosis. Colonization of trachea, OPH, and dental plaque by potential respiratory pathogens (PRPs) as Staphylococcus aureus, Pseudomonas, Klebsiella, Proteus, Acinetobacter and E. coli species was identified by culturing of OPH swab, dental swab and endotracheal tube (ETT) aspirate on inclusion into the study and every 4 days thereafter till ICU discharge, 3 weeks of ICU stay, or death. Secondary endpoints included time to VAP and its incidence, duration of MV, ICU discharge, and mortality rate.

VAP was diagnosed when patient developed; new and/or progressive infiltrates in chest radiograph plus two or more of the following; leucocytosis ≥ 12000/mm3 or leucopenia ≤ 4000c/mm3, fever > 38oC or hypothermia < 36oC, or mucopurulent secretion as evident by gross inspection. The clinically diagnosed VAP was confirmed by quantitative endotracheal aspirate at a cut off value ≥105 colony forming unit (cfu) /ml.

ELIGIBILITY:
Inclusion Criteria:

* Mechanically ventilated

Exclusion Criteria:

* None

Ages: 2 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2007-07; Primary Completion 2008-05 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Dental plaque score - oropharyngeal colonization | 21 days

SECONDARY OUTCOMES:
ventilator associated pneumonia | 21 days
Mortality | 21 days
duration of mechanical ventilation and ICU stay | 21 days